CLINICAL TRIAL: NCT00961480
Title: A 3-Part, Open-Label, Randomized, 2-Period Crossover Study to Demonstrate the Definitive Bioequivalence After Administration of the FMI Sitagliptin/Metformin 50/500 mg, 50/850 mg and 50/1000 mg FDC Tablet and Co-administration of Corresponding Doses of Sitagliptin and Metformin as Individual Tablets
Brief Title: A Study to Demonstrate the Bioequivalence of Sitagliptin/Metformin Combination Tablets and Co-administration of Sitagliptin and Metformin as Individual Tablets (0431A-095)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0431A-095; MK0431A-095; 2009_636
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment A (Active Comparator): 50 mg sitagliptin and 500 mg metformin as individual tablets
  Interventions: Drug: sitagliptin phosphate (+) metformin hydrochloride; Drug: Comparator: metformin 500mg; Drug: Comparator: sitagliptin
- Treatment B (Experimental): sitagliptin/metformin 50 mg/500 mg tablet
  Interventions: Drug: Comparator: FMI sitagliptin / metformin 50 mg/500 mg FDC tablet
- Treatment C (Active Comparator): 50 mg sitagliptin and 1000 mg metformin as individual tablets
  Interventions: Drug: Comparator: sitagliptin; Drug: Comparator: metformin 1000 mg
- Treatment D (Experimental): sitagliptin/metformin 50 mg/1000 mg tablet
  Interventions: Drug: Comparator: FMI sitagliptin/metformin 50 mg/1000 mg FDC tablet
- Treatment E (Active Comparator): 50 mg sitagliptin and 850 mg metformin as individual tablets
  Interventions: Drug: Comparator: sitagliptin; Drug: Comparator: metformin 850 mg
- Treatment F (Experimental): sitagliptin/metformin 50 mg/850 mg tablet
  Interventions: Drug: Comparator: FMI sitagliptin/metformin 50 mg/850 mg FDC tablet

INTERVENTIONS:
Drug: sitagliptin phosphate (+) metformin hydrochloride — place holder - do not post
  Arms: Treatment A
Drug: Comparator: metformin 500mg — A single dose of metformin 500 mg tablet
  Other Names: Glucophage
  Arms: Treatment A
Drug: Comparator: sitagliptin — A single dose of 50 mg sitagliptin tablet
  Other Names: Januvia
  Arms: Treatment A; Treatment C; Treatment E
Drug: Comparator: FMI sitagliptin / metformin 50 mg/500 mg FDC tablet — A single dose of FMI sitagliptin/metformin 50 mg/500 mg FDC tablet
  Arms: Treatment B
Drug: Comparator: FMI sitagliptin/metformin 50 mg/1000 mg FDC tablet — A single dose of FMI sitagliptin/metformin 50 mg/1000 mg FDC tablet
  Arms: Treatment D
Drug: Comparator: FMI sitagliptin/metformin 50 mg/850 mg FDC tablet — A single dose of FMI sitagliptin/metformin 50 mg/850 mg FDC tablet
  Arms: Treatment F
Drug: Comparator: metformin 1000 mg — A single dose of metformin 1000 mg tablet
  Other Names: Glucophage
  Arms: Treatment C
Drug: Comparator: metformin 850 mg — A single dose of metformin 850 mg tablet
  Other Names: Glucophage
  Arms: Treatment E

SUMMARY:
A three part study to demonstrate the bioequivalence of a single dose of the Final Market Image (FMI) of sitagliptin/metformin 50/500, 50/850 and 50/1000 mg Fixed-Dose Combination (FDC) tablet and co-administration of corresponding doses of sitagliptin and metformin as individual tablets. Subject will only participate in one part, receiving treatment A and B (Part I), Treatment C and D (Part II) or Treatment E and F (Part III).

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of reproductive potential test negative for pregnancy and agree to use appropriate contraception
* Subject is in good health and is a non-smoker

Exclusion Criteria:

* Subject has a history of neoplastic disease (cancer), stroke, chronic seizures, or major neurological disorder
* Subject has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* Subject is a nursing mother
* Subject consumes excessive amounts of alcohol or caffeine
* Subject has donated blood, had surgery or participated in another clinical study within the past 4 weeks

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The area under the plasma concentration-time curve (AUC) after administration of sitagliptin/metformin (50/500; 50/850; 50/1000 mg/mg) FDC tablet and co-administration of corresponding doses of sitagliptin and metformin as individual tablets. | Up to 72 hours postdose

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) for metformin after administration of sitagliptin/metformin (50/500; 50/850, 50/1000 mg/mg) FDC tablet and co-administration of corresponding doses of sitagliptin and metformin as individual tablets. | Up to 72 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC